CLINICAL TRIAL: NCT02583984
Title: Metabolomic Study in Exhaled Breath Condensate of Thoracic Surgical Patients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201505133RINC
Record Dates: First submitted 2015-10-14; First posted 2015-10-22 (Estimated); Last update posted 2016-05-25 (Estimated); Status verified 2016-05

CONDITIONS: Acute Pulmonary Insufficiency Following Thoracic Surgery; Ventilator-associated Lung Injury
MeSH Terms: interventions — Thoracic Surgical Procedures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Exhaled breath condensate
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Thoracic Surgery with Lung Resection: General anesthesia and lung separation Thoracic Surgery with Lung Resection, such as lobectomy, segmentectomy
  Interventions: Procedure: Thoracic Surgery with Lung Resection
- Thoracic Surgery without Lung Resection: General anesthesia and lung separation Thoracic Surgery without Lung Resection, such as esophageal surgery, mediastinal surgery
  Interventions: Procedure: Thoracic Surgery without Lung Resection

INTERVENTIONS:
Procedure: Thoracic Surgery with Lung Resection — General anesthesia and lung separation Thoracic surgery with lung resection, such as lobectomy, segmentectomy
  Groups: Thoracic Surgery with Lung Resection
Procedure: Thoracic Surgery without Lung Resection — General anesthesia and lung separation Thoracic surgery without lung resection, such as esophageal surgery, mediastinal surgery
  Groups: Thoracic Surgery without Lung Resection

SUMMARY:
Acute lung injury (ALI) following thoracic surgery remains a major source of morbidity and mortality after lung resection. One-lung ventilation (OLV) is usually required in thoracic surgery. OLV is also an important predictor of postoperative ALI. Recent laboratory findings suggested that tissue hypoxemia and ischemia / reperfusion injury of the collapsed lungs during OLV is the major cause of lung injury. Exhaled Breath Condensate (EBC), which is the exhalate from breath typically collected by cooling device, contains most molecules found in the airway. Metabolomics refers to systematic and scientific study of chemical processes involving metabolites. This study will collect EBC for metabolomic analysis and aim to elucidate the biochemical reactions during one-lung ventilation and pathological mechanisms of acute lung injury following thoracic surgery.

DETAILED DESCRIPTION:
Acute lung injury (ALI) following thoracic surgery remains a major source of morbidity and mortality after lung resection. Despite the advancement in both the surgical techniques and the perioperative management, the incidence of postoperative ALI remains remarkable. Risk factors for postoperative lung injury are evident, including preoperative pulmonary function, type of surgical procedure, intraoperative fluid management, one-lung ventilation, and ventilator settings. One-lung ventilation (OLV) is usually required in thoracic surgery. OLV is also an important predictor of postoperative ALI. Recent laboratory findings suggested that tissue hypoxemia and ischemia / reperfusion injury of the collapsed lungs during OLV is the major cause of lung injury. Exhaled Breath Condensate (EBC), which is the exhalate from breath typically collected by cooling device, contains most molecules found in the airway. EBC analysis has potential applications in lung disease, such as severity of airway inflammation in asthmatic patients. Collecting EBC is simple and non-invasive, in contrast to bronchoscopy for lung biopsy or bronchoalveolar lavage. Metabolomics refers to systematic and scientific study of chemical processes involving metabolites. This study will collect EBC from thoracic surgical patients before, during, and after OLV. The investigators will perform metabolomic analysis and aim to elucidate the biochemical reactions during one-lung ventilation and pathological mechanisms of acute lung injury following thoracic surgery.

ELIGIBILITY:
Inclusion Criteria:

* Thoracic surgical patients requiring lung isolation
* Pulmonary resection: lobectomy, segmentectomy
* Esophageal surgery and no pulmonary resection
* Mediastinal surgery and no pulmonary resection

Exclusion Criteria:

* Metabolic disorder
* Metabolic syndrome
* Diabetes
* Pregnancy

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Thoracic surgical patients requiring lung isolation
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2017-03; Primary Completion 2018-03 (Estimated); Study Completion 2018-03 (Estimated)

PRIMARY OUTCOMES:
Number of participants with acute lung injury following thoracic surgery | 30 days

SECONDARY OUTCOMES:
Metabolome of exhaled breath condensate associated with lung injury in thoracic surgery | 5 hours

CONTACTS AND LOCATIONS:
Overall Officials: Ya-Jung Cheng, MD, PhD, Study Chair — National Taiwan University Hospital
Locations (1):
- Department of Anesthesiology, National Taiwan University Hospital, Taipei, Taiwan